CLINICAL TRIAL: NCT06730100
Title: Phase 2 Trial of CBX-12 for Metastatic Chemotherapy-Refractory Microsatellite Stable Colorectal Cancer
Brief Title: CBX-12 for the Treatment of Metastatic Chemotherapy-Refractory Microsatellite Stable Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no accruals
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-10048; NCI-2024-10048 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10707 (Other: UPMC Hillman Cancer Center LAO); 10707 (Other: CTEP); UM1CA186690 (NIH)
Record Dates: First submitted 2024-12-11; First posted 2024-12-12 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Mismatch Repair Proficient Colorectal Carcinoma; Refractory Mismatch Repair Proficient Colorectal Carcinoma; Stage IV Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (CBX-12) (Experimental): Patients receive CXB-12 IV over 60 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo x-rays during screening, and CT, MRI, and blood collection throughout the study and patients may undergo biopsy during screening and on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: pH Low Insertion Peptide-exatecan Conjugate CBX-12; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: pH Low Insertion Peptide-exatecan Conjugate CBX-12 — Given IV
  Other Names: Alphalex Conjugate CBX-12; Alphalex-exatecan Conjugate CBX-12; CBX 12; CBX-12; CBX12; Low pH Targeting Alphalex-exatecan Conjugate CBX-12; pHLIP-exatecan Conjugate CBX-12
Procedure: X-Ray Imaging — Undergo chest x-rays
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase II trial studies how well CBX-12 works in treating patients with microsatellite stable colorectal cancer that has spread to other parts of the body (metastatic) and is no longer responding to chemotherapy treatment (chemotherapy-refractory). The usual approach to treating colorectal cancer includes treatment with surgery, radiation, or Food and Drug Administration (FDA)-approved drugs such as trifluridine-tipiracil, bevacizumab, regorafenib, or fruquintinib. However, most metastatic colorectal patients progress through all approved treatments and eventually succumb to their disease. CBX-12 is a drug that contains a peptide (a substance that contains many amino acids [molecules that join together to form proteins]) called pHLIP, linked to an anticancer substance called exatecan. Upon administration, pHLIP gets inserted into the cellular membrane of tumor cells, delivering exatecan to kill them. Giving CBX-12 may work better than the usual approach in treating patients with metastatic chemotherapy-refractory microsatellite stable colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the clinical activity, as determined by response rate, of pH low insertion peptide-exatecan conjugate CBX-12 (CBX-12) in microsatellite stable/mismatch repair proficient (MSS/pMMR) metastatic colorectal cancer (mCRC) patients.

SECONDARY OBJECTIVES:

I. To evaluate the pharmacodynamics of CBX-12 (DDR3 and apoptosis). II. To determine the effect of CBX-12 on progression-free survival (PFS).

EXPLORATORY OBJECTIVES:

I. To evaluate the tissue and plasma pharmacokinetics (PK) of CBX-12 and free exatecan.

II. To evaluate circulating tumor deoxyribonucleic acid (DNA) (ctDNA) as a predictor for treatment response to CBX-12.

III. To evaluate the safety and tolerability of CBX-12 dosed every 21 days. IV. To evaluate biomarkers of response to CBX-12 (DNA damage response, apoptosis, SLFN11 expression, TOP1-DNA complex).

OUTLINE:

Patients receive CXB-12 intravenously (IV) over 60 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo x-rays during screening, and computed tomography (CT), magnetic resonance imaging (MRI), and blood collection throughout the study and patients may undergo biopsy during screening and on study.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for 12 months or until death.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic colorectal cancer (mCRC) that is mismatch repair proficient (pMMR) based on local testing performed in a Clinical Laboratory Improvement Act (CLIA) lab
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with CT scan, MRI, or calipers by clinical exam
* Potential trial participants should have recovered from clinically significant adverse events of their most recent therapy/intervention prior to enrollment, with no Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0 toxicity of grade 3 or higher at the time of enrollment
* Availability of archival tumor tissue at the time of patient enrollment for molecular profiling studies
* Patients must have progressed on or been intolerant to at least 2 lines of prior therapies:

  * Have progressed on or intolerant of standard therapies, including a fluoropyrimidine (5-fluorouracil or capecitabine), oxaliplatin, irinotecan, and VEGF inhibitor (bevacizumab or biosimilar).
  * If left-sided primary and RAS/RAF wild-type, then have progressed on or intolerant of EGFR inhibitor (cetuximab or panitumumab).
  * If BRAF V600 mutation, then have progressed on or intolerant of BRAF inhibitor (encorafenib).
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of CBX-12 in patients <18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8.0 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) =< 3 × institutional ULN
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression for at least 4 weeks
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* Patients are willing and able to undergo pre- and on-treatment biopsies (first 10 patients in stage 1 only)
* The effects of CBX-12 on the developing human fetus are unknown. For this reason and because topoisomerase 1 inhibitors are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 6 months after the last dose of study medication. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of CBX-12 administration
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CBX-12
* Patients with concurrent administration of medication expected to cause drug interactions with CBX-12, including strong inducers and strong inhibitors of CYP3A4/1A2 isoenzymes or sensitive substrates of CYP3A4/2B6, OATP1B1, OATP1B3, OAT1, and MATE-2k
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because CBX-12 is a topoisomerase 1 inhibitors agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CBX-12, breastfeeding should be discontinued if the mother during treatment with CBX-12 and for at least 4 months after the last dose of CBX-12. Male patients treated with CBX-12 should use effective contraception and avoid fathering a child during and up to 4 months after treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-02-17 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From registration to disease progression or death due to any cause, assessed up to 12 months
  Treatment response will be assessed using Response Evaluation Criteria in Solid Tumors version 1.1. Objective response will be defined as either complete response or partial response. Simon's 2-stage optimal design will be used.
Dose limiting toxicities (DLTs) | Baseline up to 12 months
  DLTs will be defined as any grade >= 3 non-hematologic toxicity irrespective of adequate supportive treatment, or grade >= 4 hematologic toxicity per Common Terminology Criteria for Adverse Events version 5.0 attributed as possibly, probably, or definitely related to drug. The ORR will be estimated along with the 95% confidence interval.

SECONDARY OUTCOMES:
Pharmacodynamics of CBX-12 by DDR3 and apoptosis | Baseline to 12 months
  Percent of tumor cells positive for deoxyribonucleic acid (DNA) damage marker γH2AX and percent of tumor cells positive for apoptosis marker cleaved caspase 3. Pre- and on-treatment comparisons will be made within patients who provide evaluable paired biopsies, using a paired t-test. A nonparametric method will be pursued as needed. Assuming an 80% evaluable biopsy rate out of 17 patients, we would obtain 14 evaluable pre-treatment and 14 evaluable post-treatment biopsies. Using a one-sided paired t-test at a type I error rate of 0.05, this study achieves 80% power to detect a mean paired difference of 0.6 standard deviation of differences, which is deemed to be a medium effect size (Cohen, 1992). In addition, will fit a logistic regression on objective response with increase in %γH2AX-positive tumor cells and increase in %caspase 3-positive tumor cells, separately as well as simultaneously.
Progression-free survival (PFS) | From registration to disease progression or death due to any cause, assessed up to 12 months
  PFS and OS will be estimated by the Kaplan-Meier method, along with 95% confidence regions. The median time will be estimated and compared with 5.6 months of PFS and 10.8 months (Prager et al., 2023). One-sample log-rank tests will be performed against the reference curves from Prager et al. (Prager et al., 2023).
Overall survival (OS) | From registration to disease progression or death due to any cause, assessed up to 12 months
  PFS and OS will be estimated by the Kaplan-Meier method, along with 95% confidence regions. The median time will be estimated and compared with 5.6 months of PFS and 10.8 months (Prager et al., 2023). One-sample log-rank tests will be performed against the reference curves from Prager et al. (Prager et al., 2023).

OTHER OUTCOMES:
Tissue and plasma pharmacokinetics (PK) of CBX-12 and free exatecan | From baseline to 12 months
  The maximum concentration and area under the plasma drug concentration-time curve of the plasma PK will be compared descriptively with historical data. The on-treatment tumor concentrations of free exatecan and CBX-12 will be used to calculate the free exatecan:CBX-12 ratio. The ratio of plasma free exatecan Cmax:CBX-12 Cmax will be calculated. These ratios in tumor and plasma will be compared using a two-sided paired t-test, where p<0.05 will be considered statistically significant. The ratio of free exatecan:CBX-12 from the tumor is expected to greater than the ratio of the same from plasma.
Variant allele frequencies (VAF) of tumor mutations in circulating tumor DNA (ctDNA) | Baseline and at cycle 3
  VAF change will be assessed categorically for each patient (increased or decreased at cycle 3 as compared to baseline). VAF change will be compared to objective response or non-response using the Fisher's test, where p<0.05 will be considered statistically significant
Incidence and grades of adverse events | Baseline up to 12 months
  All patients who received at least one dose of CBX-12 will be considered evaluable for safety and toxicity. Continual toxicity monitoring will be used for all patients. Toxicity names, rates, and grades will be reported descriptively
Expression of YH2AX | Baseline to 12 months
  DNA damage, apoptosis, and TOP1-DNA complex markers will be measured in pre- and post-treatment samples, and a difference (increase) in expression post-treatment will also be measured on DNA damage multiplex assay. Regression analysis will be used to determine if the increase in these three biomarkers correlates with response to CBX-12.
Expression of apoptosis protein markers | Baseline to 12 months
  DNA damage, apoptosis, and TOP1-DNA complex markers will be measured in pre- and post-treatment samples, and a difference (increase) in expression post-treatment will also be measured in Luminex assay. Regression analysis will be used to determine if the increase in these three biomarkers correlates with response to CBX-12
Expression of SLFN11 | At baseline
  On immunohistochemistry. SLFN11 tumor baseline expression will be measured in pre-treatment tumor tissue and regression analysis will be used to determine if baseline SLFN11 expression correlates with response to CBX-12.
Expression of TOP1-DNA complex | Baseline to 12 months
  DNA damage, apoptosis, and TOP1-DNA complex markers will be measured in pre- and post-treatment samples, and a difference (increase) in expression post-treatment will also be measured. Regression analysis will be used to determine if the increase in these three biomarkers correlates with response to CBX-12

CONTACTS AND LOCATIONS:
Overall Officials: Chaoyuan Kuang, Principal Investigator — UPMC Hillman Cancer Center LAO
Locations (15):
- United States (15):
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm